CLINICAL TRIAL: NCT02454556
Title: A Randomized, Multicentre, Open Label, Evaluator Blinded Study to Evaluate Safety and Efficacy of Folitime® of Gemabiotech S.A., Versus Gonal-f ® of Merck Serono, in Patients With Infertility Undergoing ART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gema Biotech S.A. (Industry)
Collaborators: QUID Quality in Drugs and Devices Latin American Consulting SRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEMFOL001
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Infertility
Keywords: Assisted reproduction technologies; Follicle stimulating hormone (FSH).
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLITIME® (Experimental): Therapy will be initiated in the early follicular phase (cycle day 2 or 3) subcutaneously at a dose of 225 IU per day, until sufficient follicular development is attained.
  Interventions: Drug: FOLITIME®
- Gonal-F® (Active Comparator): Therapy will be initiated in the early follicular phase (cycle day 2 or 3) subcutaneously at a dose of 225 IU per day, until sufficient follicular development is attained.
  Interventions: Drug: Gonal-F®

INTERVENTIONS:
Drug: FOLITIME®
  Other Names: Follitropin alfa (r-hFSH)
  Arms: FOLITIME®
Drug: Gonal-F®
  Other Names: Follitropin alfa (r-hFSH)
  Arms: Gonal-F®

SUMMARY:
This is an open-label, Phase 3, randomized, two arms, multicenter, prospective, experimental study of Folitime® (a new biosimilar formulation of r-hFSH, follitropin alfa) versus the original one (Gonal-f ®).

DETAILED DESCRIPTION:
Follitropin alfa is a human follicle stimulating hormone (FSH) preparation of recombinant DNA origin, which consists of two non-covalently linked, nonidentical glycoproteins designated as the alfa- and beta-subunits. Similar to other glycoprotein hormones, FSH has a high degree of heterogeneity due to differences in the amount and/or composition of the carbohydrate residues, particularly sialic acid. FSH, the active component of r-hFSH is the most important hormone responsible for follicular recruitment and development. In order to obtain final maturation of the follicle and ovulation in the absence of an endogenous LH surge, human chorionic gonadotropin (hCG) must be given following the administration of r-hFSH when monitoring of the patient indicates that sufficient follicular development has occurred.

Secondary endpoints to be measured by the study are

Efficacy

* Total dose of r-hFSH required,
* Number of days of r-hFSH stimulation
* Percentage of patients with need to increase or lower the dose of r-hFSH,
* Number of treatment cycle cancellations and their reason
* Fertilization rate
* Number of fertilized oocytes
* Number of good quality embryos
* Number of embryos transferred
* Implantation Rate
* Biochemical pregnancy
* Clinical pregnancy 10 weeks post embryo transfer
* Pregnancy outcome

Safety

Incidence of

* OHSS (and its severity)
* Local reactions (pain, bruising, redness, itching, swelling)
* Systemic drug adverse events

Tolerability

* Frequency of patients who withdraw the study drug due to lack of tolerance
* Frequency of patients who withdraw the study drug treatment due to any reason
* Patient Reported Pain: measured by a Patients Visual Analog Scale (VAS)

Immunogenicity Measurement of possible antibodies against exogenous r-hFSH will be evaluated. Pharmacodynamics

* Number and size distribution of follicles during treatment
* Number and size distribution of follicles at the day of ovulation induction (uHCG)
* Number of follicles >14 mm on the day of hCG injection.
* Hormone parameters: serum levels of estradiol, luteinizing hormone and progesterone on the day of hCG injection
* Metaphase II oocytes;
* Number of good quality oocytes

ELIGIBILITY:
Inclusion Criteria:

* 18 to 38 years of age
* Indication for controlled ovarian stimulation and IVF or intracytoplasmic sperm injection (ICSI)
* Regular menstrual cycles (25-35 days)
* History of a maximum of two fresh cycle treatments in the present series of assisted reproductive technologies (ART) at the day of first screening (thawed cycles are not subject to that criteria)
* Body mass index (BMI) ≥18 and ≤32 kg/m2
* Basal FSH <10 IU/L (cycle day 2-5)
* Antral follicle count (AFC) ≥8 to ≤18 follicles with a diameter of <10mm (sum of both ovaries) as measured on ultrasound (US) in the early follicular phase (day 1 of the stimulation cycle or of the last cycle previous to the treatment)
* Documented history of infertility due to any of the following factors: tubal factor, male factor, unexplained infertility
* Presence of both ovaries by ultrasonography and normal uterine cavity or abnormal uterine cavity without clinical significance according to the investigator's opinion (confirmed by hysterosalpingography, saline infusion sonography or hysteroscopy within 12 months before randomization) and normal uterine cavity by transvaginal ultrasound within 3 months of treatment
* Male partner with semen analysis that is at least adequate for ICSI within 6 months prior to patient beginning down-regulation (invasive or surgical sperm retrieval, donor and/or cryopreserved sperm may be used)
* Willingness to participate in the study and to comply with the study protocol
* Signed informed consent prior to screening

Exclusion Criteria:

* Presence of pregnancy
* History of or active polycystic ovary syndrome (PCOS)
* AFC >18 follicles with a diameter of <10 mm (both ovaries combined) as measured on US in the early follicular phase (menstrual cycle day 2-5) or during
* History of >2 unsuccessful fresh ART retrieval cycles
* History of poor response to gonadotropin treatment (defined as fewer than 5 oocytes retrieved in a previous attempt)
* Any hormonal treatment within 1 month before the start of the FSH treatment, with the exception of levothyroxine)
* Egg donor
* Intrauterine leiomyomas ≥5 cm or otherwise clinically relevant pathology that could impair embryo implantation or pregnancy continuation
* Previous history of OHSS
* Ovarian cyst or enlargement of undetermined origin
* History of recurrent spontaneous abortion (3 or more, even when unexplained)
* Presence of endometriosis or hydrosalpinx
* Neoplasia, including tumors of the hypothalamus and pituitary gland
* Abnormal genital bleeding of undetermined origin
* History of extrauterine pregnancy in the previous 3 months
* Sex hormone dependent tumors of the reproductive tract and accessory organs.
* Uncontrolled thyroid or adrenal dysfunction or presence of uncontrolled endocrine disorder
* Known allergy or hypersensitivity to FSH preparations or one of their excipients or progesterone or to any of the excipients of the additional study medications
* Clinically significant abnormal findings at Visit 1 that, in the opinion of the investigator, can affect trial resulkts or subject's safety
* Administration of other investigational products within the previous month or concomitant participation in another study protocol

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Pasqualini, MD, Principal Investigator — Halitus Instituto Medico
Locations (1):
- Halitus Instituto Médico, Buenos Aires, Buenos Aires F.D., Argentina